CLINICAL TRIAL: NCT06928519
Title: Efficacy and Safety of Entacapone Combined With Madopar in the Treatment of Early Parkinson's Disease: An Observational, Multicenter, Case-Control Study
Status: Recruiting | Type: Observational
Sponsor: Yousheng Xiao (Other)
Collaborators: Jiangbin Hospital of Guangxi Zhuang Autonomous Region (Unknown); Guangxi International Zhuang Medicine Hospital (Unknown); Ethnic Hospital of Guangxi Zhuang Autonomous Region (Unknown); Guangxi Hospital Division of The First Affiliated Hospital, Sun Yat-sen University (Unknown)
Responsible Party: Sponsor-Investigator, Yousheng Xiao, Professor and Chief Physician, Department of Neurology, The First Affiliated Hospital of Guangxi Medical University, Guangxi Medical University
Organization: Guangxi Medical University (Other)
Other Study IDs: EMPD-001
Record Dates: First submitted 2025-03-22; First posted 2025-04-15 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease (PD)
Keywords: Parkinson Disease; Levodopa; Benserazide; Entacapone
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Madopar Group: Participants in this group will receive Madopar (levodopa/benserazide) as part of their routine clinical treatment. Treatment decisions, including dosage and frequency, will be made by the treating physician according to the patient's clinical condition. The typical treatment for levodopa-naïve patients is Madopar 100/25 mg taken three times daily (TID) for 24 weeks. For patients already on levodopa therapy, the physician may continue the current Madopar dosage as part of routine care. This is an observational study, and no specific interventions are assigned by the study.
- Entacapone + Madopar Group: Participants in this group will receive Entacapone (200 mg) in combination with Madopar (levodopa/benserazide, typically 100/25 mg) as part of their routine clinical treatment. The typical regimen is Entacapone 200 mg administered three times daily (TID), or at a frequency matching the patient's levodopa dosing schedule, as determined by the treating physician based on the patient's clinical condition. The study is observational in nature, and no specific intervention is assigned by the study team. All treatment decisions, including drug type, dosage, and frequency, are made by the treating physician as part of routine care.

SUMMARY:
This observational, multicenter, case-control study aims to evaluate the efficacy and safety of Entacapone combined with Madopar (levodopa/benserazide) in the treatment of early-stage Parkinson's disease (PD) among Chinese patients. The study will enroll patients diagnosed with PD according to the MDS criteria, aged 18-80, with modified Hoehn-Yahr stages 1-2.5, and who have not previously used Entacapone. Participants will be assigned to two groups based on their prior treatment history: the LBE group (levodopa/benserazide/entacapone) or the LB group (levodopa/benserazide only), according to their actual clinical treatment plan.

The study will observe patients over a 24-week period, evaluating changes in motor symptoms using the MDS-UPDRS Part III score as the primary endpoint. Secondary outcomes include assessments of daily living abilities, motor complications, quality of life (PDQ-39), cognitive function (MMSE), global impression (CGI), and safety profiles, including adverse event reporting.

This study does not involve any interventional treatment changes; all therapeutic decisions remain at the discretion of the treating physicians. The findings are expected to provide real-world evidence regarding the potential benefits and safety of adding Entacapone to Madopar in the management of early PD.

DETAILED DESCRIPTION:
This is an observational, multicenter, case-control study designed to evaluate the efficacy and safety of Entacapone combined with Madopar (Levodopa/Benserazide, LB) in the treatment of early-stage Parkinson's disease (PD) in Chinese patients. The study is conducted across multiple centers in China and includes patients diagnosed with PD according to the MDS criteria, aged 18-80 years, with a modified Hoehn-Yahr stage of 1-2.5. Participants will be divided into two groups based on their actual clinical treatment: (1) the LBE group (Levodopa/Benserazide/Entacapone) and (2) the LB group (Levodopa/Benserazide only). The study does not involve any randomization, blinding, or intervention allocation; instead, it reflects real-world clinical practice, where all treatment decisions are made solely by the attending physician.

The study will observe patients over a 24-week period to compare the effectiveness of the two treatment strategies in improving motor symptoms, daily living activities, and quality of life, as well as the incidence of adverse events. The primary outcome measure is the change in MDS-UPDRS Part III (motor examination) score from baseline to Week 24. Secondary outcomes include changes in MDS-UPDRS Part II (activities of daily living), Part IV (motor complications), total MDS-UPDRS II+III scores, PDQ-39 quality of life scores, Clinical Global Impression (CGI) scores, MMSE cognitive scores, and modified Hoehn-Yahr staging. Safety assessments include adverse events, serious adverse events, vital signs, laboratory tests, and ECG findings.

All treatments, including medication selection, dosage, and adjustment, will follow the treating physician's routine clinical judgment, and no intervention or modification by the study team will occur. Concomitant medications such as amantadine, anticholinergics, dopamine agonists, and MAO-B inhibitors (e.g., selegiline, rasagiline) are allowed if their doses are stable for at least 30 days before enrollment and remain unchanged throughout the study period.

The estimated sample size is 216 participants, with approximately 108 in each group, allowing for a 10% dropout rate. The study is expected to start in June 2025 and complete by April 2027, with final data analysis by June 2027. The results of this study aim to provide real-world evidence regarding the potential benefits and safety of Entacapone combined with Madopar in the early-stage PD population in China.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 80 years;

Diagnosed with Parkinson's Disease based on the MDS criteria, confirmed by a movement disorder neurologist;

Modified Hoehn and Yahr stage between 1 and 2.5;

No prior use of entacapone;

MMSE score ≥ 26;

BDI (Beck Depression Inventory) score < 15;

Either:

Has never used levodopa before, or

Has been on a stable dose of levodopa (300-600 mg/day) for at least 1 month prior to enrollment;

Stable doses of amantadine, anticholinergics, dopamine agonists, selegiline, or rasagiline are allowed if maintained for at least 30 days prior to and during the study;

Willing and able to give informed consent and comply with study procedures, with caregiver support if needed.

Exclusion Criteria:

Previous use of entacapone or tolcapone for more than 30 days, or within 4 weeks before baseline;

Use of dopamine agonists within 4 weeks before baseline;

BDI score ≥ 15;

MMSE score < 26;

Unstable levodopa dosage;

History of dyskinesia;

Diagnosis of atypical or secondary parkinsonism, or history of PD-related neurosurgery;

Clinically significant medical conditions within the past 5 years that could interfere with study participation;

Use of medications known to induce parkinsonism;

Participation in other investigational drug trials within 30 days before baseline.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll adult patients diagnosed with Parkinson's disease according to MDS criteria, aged between 18 and 80 years, and in the early stages of the disease (modified Hoehn-Yahr stage 1-2.5). Participants must have a Mini-Mental State Examination (MMSE) score ≥26 and a Beck Depression Inventory (BDI) score <15. Eligible patients will include those who are either levodopa-naïve or have been on a stable dose of levodopa (300-600 mg/day) for at least one month. All participants must voluntarily agree to join the study, provide informed consent, and be able to comply with the study protocol.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to Week 24 in the MDS-UPDRS Part III (Motor Examination) score | Baseline to Week 24
  The MDS-UPDRS Part III (Motor Examination) assesses the motor function of patients with Parkinson's disease. The total score ranges from 0 to 132, with higher scores indicating greater motor impairment. The change from baseline to Week 24 will be analyzed to evaluate treatment efficacy.

SECONDARY OUTCOMES:
Change from baseline to Week 24 in the MDS-UPDRS Parts II and III total score | Baseline to Week 24
  he MDS-UPDRS Part II assesses activities of daily living (maximum score: 52) and Part III assesses motor function (maximum score: 132). The combined total score (range: 0-184) reflects overall functional impairment, with higher scores indicating greater disability.
Change from baseline to Week 24 in the MDS-UPDRS Part II (Activities of Daily Living) score | Baseline to Week 24
  The MDS-UPDRS Part II evaluates the impact of Parkinson's disease on activities of daily living (ADL), such as speech, handwriting, dressing, and walking. The total score ranges from 0 to 52, with higher scores indicating greater disability. The score change from baseline to Week 24 will be analyzed to assess treatment effectiveness on daily functioning.
Change from baseline to Week 24 in the MDS-UPDRS Part IV score | Baseline to Week 24
  The MDS-UPDRS Part IV evaluates motor complications including dyskinesia and wearing-off phenomena. Changes in the score from baseline to Week 24 will be analyzed to assess treatment-related motor complications.
Change from baseline to Week 24 in the PDQ-39 summary index score | Baseline to Week 24
  The Parkinson's Disease Questionnaire-39 (PDQ-39) assesses health-related quality of life across 8 domains. The summary index score reflects the overall impact of Parkinson's disease on quality of life, with higher scores indicating worse outcomes.
Change from baseline to Week 24 in the Clinical Global Impression (CGI) score | Baseline to Week 24
  The Clinical Global Impression (CGI) scale is used by both investigators and participants to rate overall disease severity and clinical improvement. The score change from baseline to Week 24 will be used to assess perceived treatment effectiveness.
Change in modified Hoehn-Yahr stage from baseline to Week 24 | Baseline to Week 24
  The modified Hoehn-Yahr staging scale evaluates the severity and progression of Parkinson's disease, with higher stages indicating more advanced disease. Stage change from baseline to Week 24 will be used to assess disease progression or stability.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guanxi, China

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) is currently under review and will depend on ethical approvals, data use agreements, and institutional policy.

REFERENCES:
- [Background] Stocchi F, Rascol O, Kieburtz K, Poewe W, Jankovic J, Tolosa E, Barone P, Lang AE, Olanow CW. Initiating levodopa/carbidopa therapy with and without entacapone in early Parkinson disease: the STRIDE-PD study. Ann Neurol. 2010 Jul;68(1):18-27. doi: 10.1002/ana.22060. PMID 20582993
- [Background] Fung VS, Herawati L, Wan Y; Movement Disorder Society of Australia Clinical Research and Trials Group; QUEST-AP Study Group. Quality of life in early Parkinson's disease treated with levodopa/carbidopa/entacapone. Mov Disord. 2009 Jan 15;24(1):25-31. doi: 10.1002/mds.21878. PMID 18846551
- [Background] Lew MF, Somogyi M, McCague K, Welsh M; Lce QoL Study Group. Immediate versus delayed switch from levodopa/carbidopa to levodopa/carbidopa/entacapone: effects on motor function and quality of life in patients with Parkinson's disease with end-of-dose wearing off. Int J Neurosci. 2011 Nov;121(11):605-13. doi: 10.3109/00207454.2011.598982. Epub 2011 Aug 16. PMID 21843110
- [Background] Tolosa E, Hernandez B, Linazasoro G, Lopez-Lozano JJ, Mir P, Marey J, Kulisevsky J. Efficacy of levodopa/carbidopa/entacapone versus levodopa/carbidopa in patients with early Parkinson's disease experiencing mild wearing-off: a randomised, double-blind trial. J Neural Transm (Vienna). 2014 Apr;121(4):357-66. doi: 10.1007/s00702-013-1114-x. Epub 2013 Nov 20. PMID 24253234
- [Background] Hauser RA, Panisset M, Abbruzzese G, Mancione L, Dronamraju N, Kakarieka A; FIRST-STEP Study Group. Double-blind trial of levodopa/carbidopa/entacapone versus levodopa/carbidopa in early Parkinson's disease. Mov Disord. 2009 Mar 15;24(4):541-50. doi: 10.1002/mds.22343. PMID 19058133
- [Background] Liao X, Wu N, Liu D, Shuai B, Li S, Li K. Levodopa/carbidopa/entacapone for the treatment of early Parkinson's disease: a meta-analysis. Neurol Sci. 2020 Aug;41(8):2045-2054. doi: 10.1007/s10072-020-04303-x. Epub 2020 Mar 11. PMID 32162166
- [Background] Kuoppamaki M, Leinonen M, Poewe W. Efficacy and safety of entacapone in levodopa/carbidopa versus levodopa/benserazide treated Parkinson's disease patients with wearing-off. J Neural Transm (Vienna). 2015 Dec;122(12):1709-14. doi: 10.1007/s00702-015-1449-6. Epub 2015 Sep 7. PMID 26347184
- See also: Entacapone combined with levodopa/benserazide or levodopa/carbidopa in early Parkinson's disease. — https://pubmed.ncbi.nlm.nih.gov/